CLINICAL TRIAL: NCT01256515
Title: Health Management Training to Enhance Influenza Vaccine Immunogenicity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, John W. Denninger, MD, PhD, Director of Research, Benson-Henry Institute, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2009P001437; 5R01DP000339 (NIH)
Record Dates: First submitted 2010-12-07; First posted 2010-12-08 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: No Conditions
Keywords: Healthy adults aged 50 or older

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Health Education Training Group 1 (Experimental): One form of health education training
  Interventions: Behavioral: Health Education; Behavioral: Health Education Training
- Health Education Training Group 2 (Active Comparator): Another form of health education training
  Interventions: Behavioral: Health Education; Behavioral: Health Education Training

INTERVENTIONS:
Behavioral: Health Education — CDs, techniques, advice, and group training pertaining to a healthier lifestyle. Both groups will have this intervention, but the specific type of health education training will vary between groups.
Behavioral: Health Education Training — 8 weeks of group training regarding health education techniques.

SUMMARY:
The goal of this study is to assess the immunogenicity of inactivated influenza vaccination (IIV) in healthy elderly volunteers aged 50 years and older receiving one of two different health management trainings.

DETAILED DESCRIPTION:
We will obtain preliminary data on the time it takes to achieve a protective immune response, durability of response and occurrence of influenza in the following influenza season. Promising results in this age group will provide preliminary data for expanded future studies in the elderly.

ELIGIBILITY:
General Inclusion criteria are the following:

* age 50 years or older
* Infectious Disease tests - negative HIV test; hepatitis B surface antigen; anti-hepatitis C virus (HCV)
* Routine Laboratory tests
* able and willing to complete the informed consent process
* able and willing to participate for the planned duration of the study, including availability for follow-up telephone contact

General Exclusion criteria

* self report of any medical conditions for which the Center for Disease Control (CDC) states should not be vaccinated with IIV
* self-reported vaccination with the seasonal influenza vaccine for the current 2010-2011 influenza season (vaccination with the H1N1 influenza vaccine before, during, or after the study will not be exclusionary)
* history of hypersensitivity to any influenza vaccine components including thimerosal or egg
* history of Guillain-Barre syndrome
* self-reported treatment with immunomodulator/immunosuppressive drugs (interleukins (IL), corticosteroids (oral or inhaled)), G(M)- cerebrospinal fluid (CSF)) in 4 weeks before enrollment or self reported history of IL-2 administration within 5 years
* self-reported use of theophylline preparations or warfarin because of the theoretical possibilities of enhanced drug effects and toxicities following influenza vaccination
* any clinically significant abnormalities found during a routine physical examination
* self-reported history of any autoimmune disease
* acute febrile illness on the day of intended immunization - immunization deferred until illness resolved
* self report of current alcohol, substance abuse, or systemic/psychiatric illness that potentially could interfere with compliance and ability to make study visits (such as severe attention deficit hyperactivity disorder (ADHD) and current major depressive episode)

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-11; Primary Completion 2011-09 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Immunoglobin antibody response | pre and post following 8 weeks of health management training

CONTACTS AND LOCATIONS:
Overall Officials: John Denninger, M.D., Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Benson-Henry Institute, 151 Merrimac St, 4th Floor, Boston, Massachusetts, United States